## CONSENT TO ACT AS A PARTICIPANT IN A RESEARCH STUDY

**TITLE:** Open Label Study to evaluate Efficacy and Safety of Short-Term, Adjunctive Adrenocorticotropic Hormone (ACTH) Gel Therapy in Rheumatoid Arthritis

Document Date: 04/Jun/2020

Clinical Trials.gov: NCT02030028

## University of Pittsburgh

#### School of Medicine Department of Medicine

Division of Rheumatology and Clinical Immunology

#### CONSENT TO ACT AS A PARTICIPANT IN A RESEARCH STUDY

**TITLE:** Open Label Study to evaluate Efficacy and Safety of Short-Term, Adjunctive Adrenocorticotropic Hormone (ACTH) Gel Therapy in Rheumatoid Arthritis

Principal Investigator: Dana Ascherman, MD

200 Lothrop Street

Biomedical Science Tower, S723

Pittsburgh, PA 15261

24 Hour Emergency Contact Number: 412-647-7243/ pager # 2261

Co-Investigators: Larry Moreland, MD

Thaddeus Osial, MD Alan Berg, MD

Yong Gil Hwang, MD Kimberly Liang, MD Kenneth Gold MD

**Source of Support:** Questor Pharmaceuticals, Inc.

It is very important that you read and understand the following information. Please feel free to ask the study doctor or the research staff any questions that will help you understand the study and what you are expected to do. Before you agree to take part in this study, you may take this information home and discuss it with a family member or your family doctor.

#### Why is this research being done?

The purpose of this research study is to evaluate if the study drug, ACTH Gel helps decrease the disease symptoms in people with Rheumatoid Arthritis (RA) who are already taking medications prescribed by their physician and are still experiencing disease symptoms.

ACTH gel has been a Food and Drug Administration-approved treatment for Rheumatoid Arthritis since 1952, and in 2010 the FDA retained RA as a disease approved for ACTH gel use. Despite its FDA approval there is very limited data on its how well ACTH gel works in improving the symptoms of people with RA.

#### Who is being asked to take part in this research study?

You are being asked to participate in this study because you have Rheumatoid Arthritis (RA) and because you have been taking medicine prescribed by your doctor to improve your RA for at least six months but you are still having difficulty with disease symptoms. You may still have tender or swollen joints or your clinical blood tests might show that you still have inflammation (swelling) that indicates your disease is not under control.

### What procedures will be performed for research purposes?

Before any study procedures are done the study doctor and research staff will explain the study to you and ask you to read the consent form. They will answer any questions you may have about the study and what you are being asked to do. If you decide to participate you will be asked to sign this consent form and a copy will be given to you.

This study will last a total of four months from the screening visit to the last study visit. You will have a screening visit and a baseline visit. You will then be seen at two and four weeks after your baseline visit, then monthly after that until month four. Each study visit will last approximately 30 minutes and you will see the study physician and the study nurse (research coordinator) at each visit. The study visits will take place where you normally see your doctor.

What you will do at each study visit is describe below:

### **SCREENING VISIT:**

You will discuss the study thoroughly with the study doctor and the study nurse (research coordinator). You will be given the opportunity to ask questions and your questions will be answered to your satisfaction. Then you will be asked to sign this informed consent document and a copy of the signed document will be provided to you.

We will obtain a medical history from you about your RA and we will ask you about your current RA medications. The study doctor will give you a limited physical exam, focusing on your RA symptoms that includes an assessment of your tender and swollen joints. The joint exam may be performed by the study nurse. The doctor may also ask you about the impact of your disease on your daily life. We will obtain routine clinical blood from you for a Complete Blood Count, Glucose levels, Creatinine and ALT (liver function), Sedimentation Rate, and C - reactive protein. These are blood tests your doctor would order normally to see how well you are doing and to see if you have any inflammation (swelling) in your body. These tests are considered standard of care for people with Rheumatoid Arthritis and you or your insurance will be responsible for them.

If you are a female of child bearing age, we will ask you to take a urine pregnancy test at each study visit. You will not be required to perform this test at home, however the risks of taking ACTH gel, the study medication, while pregnant are unknown so we would ask that you do not become pregnant while on this study. If you are pregnant or you become pregnant during this study, you cannot participate. The only certain way to prevent pregnancy is to avoid sexual activity, however if you are using an appropriate method of birth control such as a female diaphragm, intrauterine device, or contraceptive sponge along with a male use of a condom, birth control pills, injections or implants and do not become pregnant you will be allowed to continue. The Screening visit will take about 30 minutes to complete

#### **BASELINE VISIT:**

The study doctor will give you a limited physical exam, focusing on your RA symptoms, your joint pain and/ or tenderness and your ability to perform normal tasks. The joint exam may be performed by the study nurse. You will be asked to complete a brief questionnaire describing your level activity and the impact your disease has on your ability perform daily tasks. If you are a female of child bearing age, we will ask you to take a urine pregnancy test before we give you any medication. We will obtain blood from you in the amount of 2 tablespoons for research purposes. These are not routine tests that your doctor would order and you will not know the results of these tests. You and/ or your insurance carrier will NOT be responsible for these tests.

The study nurse will teach you how to give yourself a subcutaneous (under the skin) injection. You will be asked to perform this task while the nurse is watching to make sure that you are able to this correctly at home. You will be given enough medication at this visit to last for four weeks. The dose of the study medication is 80 units given under the skin twice each week. You will be asked to complete a medication diary to document that you are taking the medication as prescribed. The study nurse will give you this diary and show you how to complete it correctly. You will also be given a sharps container to dispose of your used syringes. You will be asked to bring the sealed container to your next study visit for the research team to properly dispose of. You will be given a new sharps container at each study visit. The baseline study visit will take about 30 minutes to complete.

#### WEEK 2:

The study doctor will give you a limited physical exam, focusing on your RA symptom , your joint pain and/ or tenderness and your ability to perform normal tasks. The joint exam may be performed by the study nurse. You will be asked to complete a brief questionnaire describing your level activity and the impact your disease has on your ability perform daily tasks. We will obtain routine clinical blood from you for a Complete Blood Count, Glucose levels, Creatinine and ALT (liver function), Sedimentation Rate, and C - reactive protein. These are blood tests your doctor would order normally to see how well you are doing and to see if you have any inflammation (swelling) in your body. These tests are considered standard of care for people with Rheumatoid Arthritis and you or your insurance will be responsible for them We will obtain blood from you in the amount of 2 tablespoons for research purposes. These are not routine tests that your doctor would order and you will not know the results of these tests. You and/ or your insurance carrier will NOT be responsible for these tests.

The study nurse will ask you about any problems you have had giving yourself the medication and will ask you experienced any side effects. If you are having difficulty giving yourself the medication, the study nurse will review the injection procedure again with you. The study nurse will also ask about any other illness you may have had while taking the study medication. The Week 2 visit will take about 30 minutes to complete.

#### WEEK 4, WEEK 8, AND WEEK 12:

The study doctor will give you a limited physical exam, focusing on your RA symptoms, your joint pain and/ or tenderness and your ability to perform normal tasks. The joint exam may be performed by the study nurse. You will be asked to complete a brief questionnaire describing your level activity and the impact your disease has on your ability perform daily tasks. We will obtain routine clinical blood from you for a Complete Blood Count, Glucose levels, Creatinine and ALT (liver function), Sedimentation Rate, and C-Reactive Protein. These are blood tests your doctor would order normally to see how well you are doing and to see if you have any inflammation (swelling) in your body. These tests are considered standard of care for people with Rheumatoid Arthritis and you or your insurance will be responsible for them. We will obtain blood from you in the amount of 2 tablespoons for research purposes. These are not routine tests that your doctor would order and you will not know the results of these tests. You and/ or your insurance carrier will NOT be responsible for these tests.

The study nurse will ask you about any problems you have had giving yourself the medication and will ask you experienced any side effects. The study nurse will also ask about any other illness you may have had while taking the study medication.

You will be given enough medication at these visits to last for four weeks. You will be asked to return your completed medication diary and your sharps container with used syringes. You will be given a new medication diary to complete. You will also be given a sharps container to dispose of your used syringes. You will be asked to bring the sealed container to your next study visit for the research team to properly dispose of. You will be given a new sharps container at each study visit. These study visits will take about 30 minutes to complete.

#### WEEK 16 - FINAL STUDY VISIT:

The study doctor will give you a limited physical exam, focusing on your RA symptoms, your joint pain and/ or tenderness and your ability to perform normal tasks. The joint exam may be performed by the study nurse. You will be asked to complete a brief questionnaire describing your level activity and the impact your disease has on your ability perform daily tasks. We will obtain routine clinical blood from you for a Complete Blood Count, Glucose levels, Creatinine and ALT (liver function), Sedimentation Rate, and C-Reactive Protein. These are blood tests your doctor would order normally to see how well you are doing and to see if you have any inflammation (swelling) in your body. These tests are considered standard of care for people with Rheumatoid Arthritis and you or your insurance will be responsible for them . We will obtain blood from you in the amount of 2 tablespoons for research purposes. These are not routine tests that your doctor would order and you will not know the results of these tests. You and/ or your insurance carrier will NOT be responsible for these tests.

The study nurse will ask you about any problems you have had giving yourself the medication and will ask you experienced any side effects. The study nurse will also ask about any other illness you may have had while taking the study medication.

What are the possible risks, side effects, and discomforts of this research study?

#### Risks of the Study Drug:

ACTH gel may cause side effects similar to side effects that happen due to treatment with steroid medicines. Not all of these side effects have occurred with ACTH gel but they may occur. ACTH gel has been used in the clinical setting for many years; however, if any new risks arise, you will be informed of any significant new findings.

Risks associated with the study drug include the following:

#### Likely

- Increased blood pressure, salt, and water retention or imbalance: ACTH gel can cause increases in blood pressure, salt, and water retention, and increased elimination of potassium and calcium (minerals essential to your health). Dietary salt restriction and potassium supplementation may be necessary. Please let your doctor know if you have high blood pressure (hypertension), congestive heart failure, or kidney disease.
- Masking of symptoms of other underlying or ongoing disease or disorders: ACTH
  gel may make other diseases less likely to be diagnosed. Your doctor should monitor
  you carefully during and for a period of time following discontinuation of study drug for

signs of infection, abnormal heart issues, high blood pressure, high levels of sugar, changes in weight, and blood in your stool.

- Behavioral and mood changes: ACTH gel may be associated with mood changes
  ranging from euphoria, insomnia, irritability, mood swings, personality changes, and
  severe depression to psychosis (loss of contact with reality). Also existing emotional
  instability or psychotic tendencies may worsen. Please let your doctor know if any of
  these occur or if you have existing conditions that may worsen while receiving study
  drug.
- Symptoms of other diseases, such as diabetes and myasthenia gravis (muscle weakness), may be worsened: ACTH gel may make some existing diseases, such as diabetes, worse. Please let your doctor know if there are any changes to other conditions or diseases.

#### Infrequent

**Infections:** There is an increased chance of new infections or reactivations of old infections that are no longer active. Please let your doctor know if you have any signs of an infection such as fever or discharge or if you have a history of latent tuberculosis.

 Adrenal and pituitary gland insufficiency (decreased activity) and a disease called Cushing's syndrome may occur after prolonged use of ACTh Gel. If you are treated with ACTH gel for a long period of time, your body may alter its ability to signal between glands known as the pituitary and adrenal glands. Let your doctor know if you have any weakness, darker areas of skin, weight loss, low blood pressure (hypotension), or abdominal pain.

Signs or symptoms of a disease known as Cushing's syndrome may occur while you are receiving study drug but generally resolve after ACTH gel is stopped. Your doctor will monitor you for signs and symptoms such as deposition of fat in characteristic sites (e.g., moon face), changes in skin color, easily bruise, weight gain, muscle weakness, high blood pressure, and high sugar levels.

The safety of immunization with any vaccine, particularly live viral vaccines while receiving ACTH Gel has not been studied. Vaccinations (immunizations) against infections like the flu, tetanus, etc., work by causing your immune system to produce antibodies (molecules that your body makes to fight things like bacteria and viruses). Because ACTH Gel works by stopping your immune system from making certain antibodies, vaccination may not be fully successful in protecting you against disease. You may also experience a potential for increased infections, so it is important to tell your doctor if you develop any signs of infection such as red skin, fever, chills and/or green or white discharge (pus) from a wound. Please consult with your doctor if you

Certain types of vaccinations should be avoided while on ACTH gel:

need any vaccinations prior to receiving them.

- Gastrointestinal (GI) perforation (ulcers) and bleeding: ACTH gel can cause stomach or intestinal (GI) bleeding or ulcers, typically with long term use. Symptoms of gastrointestinal bleeding are vomiting of blood, bloody bowel movements, or black, tarry stools. Please advise your doctor if you have a past history or experience any symptoms of GI bleeding.
- Eye (ophthalmic) effects such as cataracts, infections, and glaucoma: Prolonged use of ACTH gel may result in cataracts (clouding of the lens inside the eye which leads Page 5 of 11

- to a decrease in vision) or glaucoma (eye disease in which the optic nerve is damaged). There is an increased chance of eye infections as well. Please let your doctor know if you have any vision changes.
- Decrease in bone density (osteoporosis) in subjects with long term use of ACTH
  Gel: Long term use of ACTH gel may impact your body's bone density, otherwise known
  as osteoporosis. If you are female, please let your doctor know if you are postmenopausal. Your doctor will monitor you while you are receiving study drug.

#### Rare but serious

- Immunogenicity (increased immune responses) potential: ACTH gel may alter your body's immune system so that it produces antibodies (agents that may neutralize your natural production of ACTH or that may cause you to have an allergic reaction to the drug). Please let your doctor know if you are allergic to pigs or experience an allergic reaction after injection as ACTH gel has an enhanced effect in subjects with these diseases.
- Use in subjects with hypothyroidism (low thyroid levels) or liver disease may have increased effects of the drug: Please let your doctor know if you have liver disease or low thyroid levels. You may need additional blood tests to check liver and thyroid function.

Reproductive Risks: ACTH gel may result in death to unborn babies in the womb. There are no adequate and well-controlled studies in pregnant women. You should not get pregnant while being treated and should alert your doctor if you suspect you might be pregnant. A pregnancy test will be conducted to confirm that you are not pregnant at the beginning of this study. Avoiding sexual activity is the only certain method to prevent pregnancy. However, females of child-bearing potential must be willing to use an appropriate method of birth control (such as female use of a diaphragm, intrauterine device (IUD), or contraceptive sponge, in addition to male use of a condom) or the female should be using prescribed "birth control" pills, injections, or implants throughout the study. Even with use of these birth control measures, pregnancy could still result. The risks of receiving the study drug while pregnant include potential loss of pregnancy or possible birth defects. Females of child-bearing potential will undergo a urine pregnancy test prior to each exposure to the study drug.

### Other Risks:

There are also risks that are associated with the procedures used in this study, including:

**Venipuncture** (the process of drawing blood samples)

The risks of drawing blood include temporary discomfort from the needle stick, bruising, bleeding, fainting, and rarely, infection.

### Subcutaneous (under the skin) Injections

Injections into the skin may be less convenient than other forms of treatment such as oral medications. In addition, injections may cause momentary discomfort and other local symptoms, such as bleeding, bruising, redness, and, rarely, infection.

- Loss of privacy: Every effort will be made to protect your privacy and information will be handled in a confidential manner. The only information that will be provided with your stored blood is a study code. Files that link your name to the code number will be kept in a locked cabinet and only the study staff will have access to them. The samples will be provided to the researchers in such a manner whereby it will not be possible for them to connect your identity with the sample or medical information. Information about race, ethnicity, sex and medical history may be made available to the investigators studying the blood samples. Such information might be important for research. Although no one can absolutely guarantee confidentiality, using a code number greatly reduces the chance that someone will ever be able to link your name to your sample or to your results.
- Confidentiality: All records pertaining to your involvement in this research study will be stored in locked file cabinets. Only a subject number in these records will identify you. Any information about your participation in this study will be handled in a confidential manner consistent with other identifiable health information. You will not be specifically identified in any publication of research results.
- Assessment tools for Efficacy (questionnaires): You may feel uncomfortable answering
  questions about your daily activities and how your RA impacts your ability to perform daily
  tasks.

### What are the potential benefits from taking part in this research study?

A possible benefit of this study may be an improvement in your disease symptoms. However, there may be no direct benefit to participants in this study. There is no guarantee that you will receive any personal benefit from participating in this research study. It is hoped that the information gained from the study will be beneficial to patients in the future. Because of your participation, there may be advancement in knowledge about Rheumatoid Arthritis and responses to Acthar Gel drug administration.

## What treatment or procedures are available if I decide not to take part in this research study?

You do not have to participate in this study to receive treatment for your condition. The study drug, ACTH gel, offered in this study is in addition to the medications your doctor has currently prescribed for you. If you decide not to take part in this study or are withdrawn from the study, you have the option of having your personal doctor manage your disease using available drugs or treatments. The study doctor will discuss these alternative options with you.

## If I agree to take part in this research study, will I be told of any new risks that may be found during the course of the study?

You will be promptly notified if any new information (either good or bad) develops during the conduct of this research study which may cause you to change your mind about continuing to participate. If new information is provided to you, your consent to continue participation in this study will be re-obtained.

#### Will I be paid to participate in this study?

You will NOT be paid to participate in this study. We will provide you with \$50.00 at the completion of each study visit to help cover the costs of travel and/ or lost wages. We will also provide you with complimentary parking.

## Will I or my insurance provider be charged for the costs of any procedures performed as part of this research study?

You or your insurance will not be billed for any research procedures conducted as part of this study. The study drug, Acthar Gel will be provided by Questcor Pharmaceutical, Inc. and there will be no cost to you for the study drug. You and/or your insurance will be billed for standard of care costs (not study related) like the routine clinical blood tests or emergent care that you receive and you will be responsible for costs not covered by your insurance provider. You will be responsible for any applicable co-pays, co-insurances, and deductibles.

Who will pay if I am injured as a result of taking part in this research study? University of Pittsburgh researchers and their associates who provide services at UPMC recognize the importance of your voluntary participation in their research studies. These individuals and their staff will make reasonable efforts to minimize, control, and treat any injuries that may arise as a result of this research. If you believe that you are injured as a result of the research procedures being performed, please contact immediately the Principal Investigator listed on the first page of this form.

Emergency medical treatment for injuries solely and directly related to your participation in this research study will be provided to you by the hospitals of UPMC. It is possible that that UPMC may bill your insurance provider for the costs of this emergency treatment, but none of these costs will be charged directly to you. If your research-related injury requires medical care beyond this emergency treatment, you will be responsible for the costs of this follow-up care unless otherwise specifically stated below. There is no plan for monetary compensation. You do not, however, waive any legal rights by signing this form.

### Who will know about my participation in this research study?

Any information about you obtained from or for this research will be kept as confidential (private) as possible. All records related to your involvement in this research study will be stored in locked file cabinets. Your identity on these records will be indicated by a code number rather than by your name, and the information linking these code numbers with your identity will be kept separate from the research records. You will not be identified by name in any publication of research results unless you sign a separate form giving your permission (release). The University of Pittsburgh policy requires that all research records be kept for seven years following the end of a research study.

At the end of this research study, data (information) will be permanently stored in a research consortium database at the University of Pittsburgh, so that data from different Rheumatoid Arthritis research studies can be pooled together to make stronger conclusions on how to measure the symptoms of this disease. Your identity on this research data will be indicated by a code number as indicated above. Research blood will be used for Rheumatoid Arthritis specific and associated auto antibodies. The remainder of the sample will be stored indefinitely in the research repository located at the University of Pittsburgh, Division of Rheumatology.

## Will this research study involve the use or disclosure of my identifiable medical information?

This research will involve the recording of current and/or future identifiable medical information from your hospital and/or other (e.g., physician office) records. The information that will be recorded is limited to the routine clinical blood test performed at the study visits. These results will appear in your medical record and will be recorded in your research file held at University of Pittsburgh Division of Rheumatology Offices.

## Who will have access to identifiable information related to my participation in this research study?

In addition to the investigators listed on the first page of this authorization (consent) form and their research staff, the following individuals will or may have access to identifiable information (which may include your identifiable medical information) related to your participation in this research study.

Authorized representatives of the University of Pittsburgh Research Conduct and Compliance Office may review your identifiable research information (which may include your identifiable medical information) for the purpose of monitoring the appropriate conduct of this research study.

In unusual cases, the investigators may be required to release identifiable information (which may include your identifiable medical information) related to your participation in this research study in response to an order from a court of law. If the investigators learn that you or someone with whom you are involved is in serious danger or potential harm, they will need to inform, as required by Pennsylvania law, the appropriate agencies.

Authorized representatives of the sponsor of this research study ,Questcor Pharmaceutical representatives and from the University of Pittsburgh acting as the Clinical Coordinating Center for this study will review and/or obtain identifiable information (which may include your identifiable medical information) related to your participation in this research study for the purpose of monitoring the accuracy and completeness of the research data and for performing required scientific analysis of the research data. The investigators involved in the conduct of this research study will receive funding from the sponsor to perform the research procedures and to provide identifiable research and medical information related to your participation in the study.

Authorized representatives of the U.S. Food and Drug Administration may review and/or obtain identifiable information (which may include your identifiable medical information) related to your participation in this research study for the purpose of monitoring the accuracy of the research data. While the U.S. Food and Drug Administration understands the importance of maintaining the confidentiality of your identifiable research and medical information, the University of Pittsburgh and UPMC cannot guarantee the confidentiality of this information after it has been obtained by the U.S. Food and Drug Administration.

Authorized representatives of the UPMC hospitals, Clinical and Translational Research Center (CTRC) or other affiliated health care providers may have access to identifiable information (which may include your identifiable medical information) related to your participation in this research study for the purpose of (1) fulfilling orders, made by the investigators, for hospital and health care services (e.g. diagnostic procedures) associated with research study participation; (2) addressing correct payment for tests and procedures ordered by the investigators; and/or (3) for internal hospital operations (e.g. quality assurance).

## For how long will the investigators be permitted to use and disclose identifiable information related to my participation in this research study?

The investigators may continue to use and disclose, for purposes described above, identifiable information (which may include your identifiable medical information) related to your participation in this research study for a minimum of 5 years and for as long (indefinite) as it may take to complete this research study.

## May I have access to my medical information that results from my participation in this research study?

In accordance with the UPMC Notices of Privacy Practices document that you have been provided, you are permitted access to information (including information resulting from your participation in this research study) contained within your medical records filed with your health care provider unless otherwise specifically stated below.

You agree that, while the study is still in progress, you may not be given access to medical information about you that is related to the study. While a request for access to medical information can be denied, the study doctor and staff will not automatically deny a request, but will consider whether it's medically appropriate under the circumstances to allow access. Your agreement that you may be denied access to your study-related medical information during the study will not be used to deny you access to that information after the study is completed at all locations and study results are analyzed. As previously stated you will not be permitted access to results of the blood analysis.

### Is my participation in this research study voluntary?

Your participation in this research study, to include the use and disclosure of your identifiable information for the purposes described above, is completely voluntary. (Note, however, that if you do not provide your consent for the use and disclosure of your identifiable information for the purposes described above, you will not be allowed, in general, to participate in the research study) Whether or not you provide your consent for participation in this research study will have no effect on your current or future relationship with the University of Pittsburgh. Whether or not you provide your consent for participation in this research study will have no effect on your current or future care at UPMC hospitals or affiliated health care provider or your current or future relationship with a health care insurance provider.

If your doctor is involved as an investigator in this research study, as both your doctor and a research investigator, s/he is interested both in your medical care and the conduct of this research study. Before agreeing to participate in this research study, or at any time during your study participation, you may discuss your care with another doctor who is not associated with this research study. You are not under any obligation to participate in any research study offered by your doctor.

May I withdraw, at a future date, my consent for participation in this research study? You may withdraw, at any time, your consent for participation in this research study, to include the use and disclosure of your identifiable information for the purposes described above. (Note, however, that if you withdraw your consent for the use and disclosure of your identifiable medical record information for the purposes described above, you will also be withdrawn, in general, from further participation in this research study.) Any identifiable research or medical information recorded for, or resulting from, your participation in this research study prior to the date that you formally withdrew your consent may continue to be used and disclosed by the investigators for the purposes described above.

To formally withdraw your consent for participation in this research study you should provide a written and dated notice of this decision to the principal investigator of this research study at the address listed on the first page of this form.

Your decision to withdraw your consent for participation in this research study will have no effect on your current or future relationship with the University of Pittsburgh. Your decision to withdraw your consent for participation in this research study will have no effect on your current or future medical care at UPMC hospitals or affiliated health care provider or your current or future relationship with a health care insurance provider.

# If I agree to take part in this research study, can I be removed from the study without my consent?

No guarantee is made as to the results of your participation in this study. If certain circumstances were to occur, the physician may stop the study medication and your participation in this study may be terminated without your permission. These circumstances would be related to either your failure to cooperate fully with the conduct of the study, or the recognition of significant medical risks associated with your continued participation in this study. If your participation in this study is stopped, the reasons will be discussed with you.

#### **VOLUNTARY CONSENT**

All of the above has been explained to me and all of my current questions have been answered. I understand that I am encouraged to ask questions about any aspect of this research study during the course of this study, and that such future questions will be answered by the researchers listed on the first page of this form. Any questions which I have about my rights as a research participant will be answered by the Human Subject Protection Advocate of the IRB Office, University of Pittsburgh (1-866-212-2668).

| By signing this form, I agree to participate will be given to me. | ate in this research study. | A copy of this consent form |
|---|---|---|
| Printed Name of Participant | | |
| Participant's Signature | Date | Time |

### **CERTIFICATION of INFORMED CONSENT**

I certify that I have explained the nature and purpose of this research study to the above-named individual(s), and I have discussed the potential benefits and possible risks of study participation. Any questions the individual(s) have about this study have been answered, and we will always be available to address future questions as they arise."

| Printed Name of Person Obtaining Consent | Role in Research Study |
|------------------------------------------|------------------------|
| Signature of Person Obtaining Consent | Date /Time |